CLINICAL TRIAL: NCT05515172
Title: Resilience Intervention in Times of Crisis for Health Professionals During the COVID-19 Contingency
Brief Title: Resilience Intervention for Health Professionals COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Monterrey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20191210-CEI
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Mental Health Wellness 1
Keywords: mindfulness; resilience; COVID-19; nurses
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Mindfulness-based intervention is composed of micropractices, cohesion groups, affirmations, and journaling. This was administered via a webpage designed for this intervention.
  Interventions: Other: Mindfulness-based Intervention

INTERVENTIONS:
Other: Mindfulness-based Intervention — The intervention was designed by a volunteer multidisciplinary team expert in different mind-body medicine techniques (for example, medicine, psychology, thanatology, meditation, health, and wellness coaches, certified Qi Gong, and yoga instructors) and is made up of 3 components main: "micropractices," cohesion and support groups, which will be implemented for a period of 12 weeks.

SUMMARY:
In the fight against the coronavirus (COVID-19) pandemic, health personnel, especially nursing staff, have been facing enormous pressure, including a high risk of infection and inadequate protection against contamination, overwork, frustration, discrimination, isolation, lack of contact with their families and exhaustion. Therefore, the World Health Organization (WHO) has requested particular interventions to promote emotional well-being in health workers exposed to COVID-19, which must be implemented immediately, especially those aimed at women and nursing staff. . Psychological support services, including counseling or intervention via phone, internet, and apps, have been widely deployed by local and national mental health institutions in response to the COVID-19 outbreak. Complementing these efforts, the present study seeks, through mind-body medicine strategies, to promote resilience among nurses exposed to COVID-19 in critical phases. A multidisciplinary team of expert volunteers designed the intervention in different mind-body medicine techniques (for example, medicine, psychology, thanatology, meditation, health, and wellness coaches, certified Qi Gong, and yoga instructors) and is made up of 3 components main: "micropractices," cohesion and support groups, which will be implemented for 12 weeks in health personnel. This intervention responds to the international call to promote health personnel's physical and emotional health during the COVID-19 pandemic, offering an opportunity to accompany them during this time and mitigate the effects on health in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Exclusion Criteria:

* Lack of signature in the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 371 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 6 months follow-up of Subjective Well-being | At baseline, and 6 months follow-up
  Subjective Well-Being will be measured using the PERMA Profiler which evaluates positive emotions, engagement, relationships, meaning, accomplishments, perception of health, and negative emotions.
Change from Baseline to 6 months follow-up of Negative Emotions | At baseline, and 6 months follow-up
  Negative Emotions will be measured using the PERMA Profiler which evaluates positive emotions, engagement, relationships, meaning, accomplishments, perception of health, and negative emotions.
Change from Baseline to 6 months follow-up of Perception of Health | At baseline, and 6 months follow-up
  Perception of Health will be measured using the PERMA Profiler which evaluates positive emotions, engagement, relationships, meaning, accomplishments, perception of health, and negative emotions.
Change from Baseline to 6 months follow-up of Stress | At baseline and 6 months follow-up
  Stress will be measured using the perceived stress scale.
Change from Baseline to 6 months follow-up of Resilience | At baseline and 6 months follow-up
  Resilience will be measured using the brief resilience scale
Change from Baseline to 6 months follow-up of mindfulness | At baseline and 6 months follow-up
  Resilience will be measured using the mindfulness-awareness attention scale
Change from Baseline to 6 months follow-up of burnout | At baseline and 6 months follow-up
  Burnout will be measured using the Burnout Clinical Subtypes Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- TecSalud, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cepeda-Lopez AC, Solis Dominguez L, Villarreal Zambrano S, Garza-Rodriguez IY, Del Valle AC, Quiroga-Garza A. A comparative study of well-being, resilience, mindfulness, negative emotions, stress, and burnout among nurses after an online mind-body based intervention during the first COVID-19 pandemic crisis. Front Psychol. 2023 Mar 13;14:848637. doi: 10.3389/fpsyg.2023.848637. eCollection 2023. PMID 36993886